CLINICAL TRIAL: NCT01842100
Title: To Compare the Strategies of Universal Antibiotic Prophylaxis Versus Screen-and-treat in Reducing Infective Complications and Re-infection in Women Who Undergo Termination of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QMHRC99 - 15 RC/B/121
Record Dates: First submitted 2013-04-21; First posted 2013-04-29 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Induced Abortion; Postaboral Pelvic Inflammatory Disease; Sexually Transmitted Infections
Keywords: Induced abortion; Postaboral pelvic inflammatory disease; Sexually transmitted infections; Universal antibiotic prophylaxis; Screen-and-treat approach
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Universal antibiotic prophylaxis (Active Comparator): In the universal prophylaxis group, all women received doxycycline 100 mg twice daily for 7 days starting on the day of induced abortion. Screening for sexually transmitted diseases was done as baseline but the results were not revealed to the patients.
  Interventions: Drug: Universal antibiotic prophylaxis
- Screen-and-treat (Active Comparator): In the screen-and-treat group, the results of screening for sexually transmitted infections (STI) were revealed to the patients. They would only receive appropriate specific antibiotics treatment only if they were screened positive for any of the STIs. If they were found to have STI, their sexual partners would also be referred to the local social hygiene clinics for contact tracing and treatment. Contraception by barrier methods would also be advised.
  Interventions: Other: Screen-and-treat

INTERVENTIONS:
Drug: Universal antibiotic prophylaxis — 100 mg twice daily for 7 days starting on the day of induced abortion
  Arms: Universal antibiotic prophylaxis
Other: Screen-and-treat — Specific antibiotic treatment was only given if the women was found to have sexually transmitted infection(s) on screening.
  Arms: Screen-and-treat

SUMMARY:
Screen-and-treat approach reduces postabortal pelvic inflammatory disease after induced abortion, and at the same time alters women's sexual behavior and prevents further re-infection by sexually transmitted infections when compared to the universal antibiotic prophylaxis strategy.

DETAILED DESCRIPTION:
While universal antibiotic prophylaxis during induced abortion has been proven to reduce postabortal pelvic inflammatory diseases, screen-and-treat approach has the potential benefit of altering women's sexual behavior and preventing further re-infection by sexually transmitted infections. We conducted a randomized controlled trial to compare the effect of the two approaches in preventing postabortal pelvic inflammatory disease and the women's sexual behavior.

ELIGIBILITY:
Inclusion Criteria:

* women requesting for induced abortion in the gynecology clinic

Exclusion Criteria:

* nil

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2193 (Actual)
Dates: Start 1999-09; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Rate of postabortal inflammatory disease 6 weeks after induced abortion. | 6 weeks after induced abortion.

SECONDARY OUTCOMES:
Rate of re-infection by sexually transmitted infections 24 weeks after induced abortion. | 24 weeks after induced abortion.
Proportion of women having abstinence from sexual intercourse or using condom at 6 weeks, 24 weeks and 1 year after induced abortion. | 6 weeks, 24 weeks and 1 year after induced abortion

CONTACTS AND LOCATIONS:
Overall Officials: Sofie SF Yung, MBBS, MRCOG, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, China